CLINICAL TRIAL: NCT05440682
Title: Structural and Functional Connectivity as Outcome Markers of Cranioplasty Following Decompressive Craniectomy
Brief Title: Connectivity in Cranioplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Usl di Bologna (Other Government)
Collaborators: Ministero della Salute, Italy (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISNB-MR&NR-2020-01
Record Dates: First submitted 2022-03-28; First posted 2022-07-01 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Acquired Brain Injury; Traumatic Brain Injury; Ischemic Stroke; Hemorrhagic Stroke
Keywords: Decompressive Craniectomy; Cranioplasty; MRI; EEG; Functional Connectivity; Structural Connectivity.
MeSH Terms: conditions — Brain Injuries; Brain Injuries, Traumatic; Ischemic Stroke; Hemorrhagic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CP group (Experimental): Pre- post-cranioplasty and 6 months follow-up MRI assessment. Each MRI session lasts about 60 minutes and will measure Diffusion Tensor Imaging, Tractography and resting state fMRI
  Interventions: Procedure: CP group

INTERVENTIONS:
Procedure: CP group — Pre- post-cranioplasty and 6 months follow-up MRI assessment. Each MRI session lasts about 60 minutes and will measure Diffusion Tensor Imaging, Tractography and resting state fMRI.

SUMMARY:
An Exploratory Interventional study to assess the effects of cranioplasty on brain network connectivity, neuropsychological and motor functioning in patients with severe acquired brain injury with pre-, post-cranioplasty and 6 months follow-up assessments.

DETAILED DESCRIPTION:
BACKGROUND: Cranioplasty (CP) refers to the surgical reconstruction of the cranial defect secondary to Decompressive Craniectomy (DC). The aim of this intervention is not only to restore cranial cosmesis and the normal cerebral protection, but also to facilitate neurological rehabilitation.

Clinical improvements after CP, may occur as early as 4 days after the surgical reconstruction of the cranial vault and may include vigilance/consciousness, sensorimotor and cognitive functioning. In particular, several studies showed relevant neurological improvement of motor and cognitive impairments as well as in the disability level in severe acquired brain injury (sABI) patients treated with DC in the acute phase. To date, it is not possible to predict the extent of the expected improvement after CP, and the effects in terms of long-term functional outcome appears to be variable from subject to subject.

The CO-CRAN (COnnectivity in CRANioplasty) study is based on the experimental hypothesis that the extent of recovery could be significantly correlated with the degree of integrity of the neural network, in relation to the primary damage, of the cerebral hemisphere ipsilateral to craniectomy. It is assumed that if the neural network is relatively intact, the extent of the recovery could be maximal. Conversely, when there is an extensive functional impairment of the underlying craniectomy flap, the impairment of the neural network does not allow a maximum recovery.

AIM: The aim of the study is to investigate possible morpho-functional neuroimaging determinants that may be predictive of post-cranioplasty recovery in patients with sABI undergoing DC.

METHODS: Exploratory clinical trial with pre-test, post-test, and 6 months follow-up assessments. Medical drugs and device are not involved in the study. The design provides only one group of patients who underwent CP.

POPULATION: Patients with sABI treated with DC will be recruited in the Neurorehabilitation Unit of the IRCCS Istituto delle Scienze Neurologiche di Bologna. Subjects will be recruited accordingly to the following eligibility criteria:

* Inclusion Criteria:

  1. Diagnosis of sABI, a neurological condition due to a severe acquired brain damage (i.e., traumatic brain injury, ischemic stroke, hemorrhagic stroke) with a coma lasting at least 24 hours, according to a Glasgow Coma Scale equal or lower than 8 and/or complex and severe neurological disabilities treatable only in high specialty neurehabilitative settings.
  2. Early DC, within 24 h;
  3. Age between 18 and 75 years;
  4. Intra-hospital rehabilitation setting (ordinary hospitalization or day hospithal);
  5. Informed consent agreement.
* Exclusion Criteria:

  1. Medical instability at enrollment, defined as the acute onset of an unexplained derangement of vital parameters (i.e., temperature, blood pressure, pulse rate, respiratory rate, oxygen saturation, level of responsiveness) outside the normal range (for example, fever, acute internist conditions, etc.) and/or the onset of any new medical condition requiring unexpected additional diagnostic procedures and treatments (for example, severe pain, reduction of urinary output, etc.);
  2. Post-traumatic agitation;
  3. Dehiscence, in progress, of the DC surgical wound;
  4. CP already performed;
  5. Magnetic Resonance Imaging (MRI) absolute contraindications.

INTERVENTION: 3-T MRI scanner with a 64-channel head for structural and functional imaging (Diffusion Tensor Imaging, Tractography and resting state fMRI).

CONTROL: There is no control group, although normative data relating to a population of healthy subjects, matched by sex and age, are used to define normative parameters for functional imaging.

OUTCOMES: Multidisciplinary assessment with clinical and neurophysiological indices. All of the assessment measures will be administrated following the same timing: Pre-test: within 10 days before CP; Post-test: from 30 to 40 days after CP; Follow-up: from 170 to 190 days after CP.

EXPECTED RESULTS: The Study results may inform on the correlation between neurophysiological changes in terms of structural and functional connectivity after DC and long term cognitive, motor and clinical outcomes.

RANDOMIZATION: N/A

ASSESSOR AND PATIENT BLINDNESS: N/A

CASE REPORT AND DATA MONITORING: Specific case report forms (CRF) for every clinical and motor scale in the assessments are already available and will be used. All information about neurophysiological results will be promptly reported on the electronic database. A researcher will be responsible for the electronic database, data analyses and will draft the single patient record at the end of all procedures. In case of lost to follow-up, the information available up to that moment will be considered

SAMPLE SIZE: From the retrospective analysis of hospitalizations carried out in previous years, it is estimated that the incidence of patients with DC is around 23% per year. Therefore, out of a total of about 65 annual hospitalizations, it is estimated that 10 patients can be enrolled within two years.

DATA ANALYSES: Considering the exploratory nature of the study, descriptive statistics in the pre-post and follow-up time points will be reported and compared. The analysis will be performed by one-way ANOVA for continuous variables and Mann-Witney test for ordinal variables

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of sABI, a neurological condition due to a severe acquired brain damage (i.e., traumatic brain injury, ischemic stroke, hemorrhagic stroke) with a coma lasting at least 24 hours, according to a Glasgow Coma Scale equal or lower than 8 and/or complex and severe neurological disabilities treatable only in high specialty neurehabilitative settings.
* Early DC, within 24 h;
* Age between 18 and 75 years;
* Intra-hospital rehabilitation setting (ordinary hospitalization or day hospithal);
* Informed consent agreement.

Exclusion Criteria:

* Medical instability at enrollment, defined as the acute onset of an unexplained derangement of vital parameters (i.e., temperature, blood pressure, pulse rate, respiratory rate, oxygen saturation, level of responsiveness) outside the normal range (for example, fever, acute internist conditions, etc.) and/or the onset of any new medical condition requiring unexpected additional diagnostic procedures and treatments (for example, severe pain, reduction of urinary output, etc.);
* Post-traumatic agitation;
* Dehiscence, in progress, of the DC surgical wound;
* CP already performed;
* Magnetic Resonance Imaging (MRI) absolute contraindications.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-10-27 (Actual); Primary Completion 2021-05-12 (Actual); Study Completion 2023-04-27 (Estimated)

PRIMARY OUTCOMES:
Changes in Mean Diffusivity values: | pre-test: within 10 days before CP - post-test: from 30 to 40 days after CP - follow-up: from 170 to 190 days after CP
  - Mean diffusivity (MD) from the Diffusion Tensor Imaging (DTI) data: a measure of brain structural integrity which describes the rotationally invariant magnitude of water diffusion within brain tissues. Higher values indicate worse tissue injury.

SECONDARY OUTCOMES:
Changes in fractional anisotropy values | pre-test: within 10 days before CP - post-test: from 30 to 40 days after CP - follow-up: from 170 to 190 days after CP
  - fractional anisotropy (FA) [0-1] from the Diffusion Tensor Imaging (DTI) data: a measure of brain structural integrity which reflects the directionality of molecular displacement by diffusion. Lower values indicate worse tissue injury.
Changes in Cognitive functioning | pre-test: within 10 days before CP - post-test: from 30 to 40 days after CP - follow-up: from 170 to 190 days after CP
  LCF (Levels of Cognitive Functioning) [1-10]: a single item scale that allows to monitor cognitive and behavioral evolution from coma (LCF1) to the complete social and work reintegration (LCF 10); where higher scores mean a better outcome
Changes in disability level | pre-test: within 10 days before CP - post-test: from 30 to 40 days after CP - follow-up: from 170 to 190 days after CP
  DRS (Disability Rating Scale) [29-0]: an 8 item scale (three of them by Glasgow Coma Scale) that assess clinical changes, where higher ratings indicate a more severe disability
Changes in functional independence | pre-test: within 10 days before CP - post-test: from 30 to 40 days after CP - follow-up: from 170 to 190 days after CP
  FIM (Functional Independence Measure) [18-126]: to assess cognitive and motor abilities, where higher scores mean a better outcome
Changes in level of consciousness | pre-test: within 10 days before CP - post-test: from 30 to 40 days after CP - follow-up: from 170 to 190 days after CP
  CRS-R (Coma Recovery Scale Revised) [0-29]: to measure the behavioral correlates of state of consciousness (in patients with LCF 1-3); higher scores indicate a better outcome
Changes in functional abilities | Frame: pre-test: within 10 days before CP - post-test: from 30 to 40 days after CP - follow-up: from 170 to 190 days after CP
  EFA (Early Functional Abilities) [12-60]:to assess cognitive and motor problems in patients with disorders of consciousness or early confusional state (in patients with LCF 1-5); higher scores indicate a better outcome.
Changes in motor abilities | pre-test: within 10 days before CP - post-test: from 30 to 40 days after CP - follow-up: from 170 to 190 days after CP
  TCT (Trunk Control Test) [0-100] for trunk control aspects; (in patients with LCF 5-10); higher scores indicate a better outcome
Changes in trunk control | pre-test: within 10 days before CP - post-test: from 30 to 40 days after CP - follow-up: from 170 to 190 days after CP
  UTAS (Unified Trunk Assessment Scale) [0-31]: for trunk control aspects; (in patients with LCF 5-10); higher scores indicate a better outcome
Changes in balance control | pre-test: within 10 days before CP - post-test: from 30 to 40 days after CP - follow-up: from 170 to 190 days after CP
  UBS (Unified Balance Scale) [0-33]: to assess balance and walk; (in patients with LCF 5-10); higher scores indicate a better outcome
Changes in Ambulation | pre-test: within 10 days before CP - post-test: from 30 to 40 days after CP - follow-up: from 170 to 190 days after CP
  FAC (Functional Ambulation Categories) [0-5], WHS [1-6] and 10 meters walking test [sec]: to assess balance and walk; (in patients with LCF 5-10); higher scores indicate a better outcome
Changes in walking handicap | pre-test: within 10 days before CP - post-test: from 30 to 40 days after CP - follow-up: from 170 to 190 days after CP
  WHS (Walking Handicap Scale) [1-6] and 10 meters walking test [sec]: to assess balance and walk; (in patients with LCF 5-10); higher scores indicate a better outcome
Changes in walking abilities | pre-test: within 10 days before CP - post-test: from 30 to 40 days after CP - follow-up: from 170 to 190 days after CP
  10 meters walking test [sec]: to assess balance and walk; (in patients with LCF 5-10); higher scores indicate a better outcome
Changes in motor autonomy | pre-test: within 10 days before CP - post-test: from 30 to 40 days after CP - follow-up: from 170 to 190 days after CP
  Barthel Index [0-100]: concerning the level of motor autonomy in the activities of daily living. Lower scores indicate a better outcome
Changes in cognitive level | pre-test: within 10 days before CP - post-test: from 30 to 40 days after CP - follow-up: from 170 to 190 days after CP
  ConfuScale [0-72]: a brief neuropsychological scale to assess cognitive functioning; (in patients with LCF 4-7); higher scores indicate a better outcome
Changes in neuropsychological functions | pre-test: within 10 days before CP - post-test: from 30 to 40 days after CP - follow-up: from 170 to 190 days after CP
  ACE-R (AddenBrooke's Cognitive Examination-Revised) [0-100]: a brief neuropsychological scale to assess cognitive functioning; (in patients with LCF 4-7); higher scores indicate a better outcome.
Changes in Structured neuropsychological assessment | pre-test: within 10 days before CP - post-test: from 30 to 40 days after CP - follow-up: from 170 to 190 days after CP
  The Extensive neuropsychological battery to test the different cognitive functions (for patients with LCF>7). A z-score greater than 0 indicates an above-average performance
Changes in quantitative EEG | Frame: pre-test: within 10 days before CP - post-test: from 30 to 40 days after CP - follow-up: from 170 to 190 days after CP
  AFR score (Amplitude Frequency Reactivity) [0-10]: A standard EEG score for basic assessment of EEG features. higher values indicate a better outcome.
Changes in EEG connectivity and continuity | pre-test: within 10 days before CP - post-test: from 30 to 40 days after CP - follow-up: from 170 to 190 days after CP
  Score of the correlation between EEG signals over the scalp electrodes [0-1]. higher scores indicate a better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs - Istituto Delle Scienze Neurologiche, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No